CLINICAL TRIAL: NCT02742142
Title: Randomized Clinical Trial on Preventing and Arresting Root Surface Caries Using Silver Diammine Fluoride Solution in Older Adults Living in Fluoridated and Non-fluoridated Areas
Brief Title: Fluoride Application on Preventing and Arresting Root Caries in Fluoridated and Non-fluoridated Areas
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UW12-296
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Water; silver diamine fluoride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Placebo Comparator): Distilled water as placebo with a bitter flavor added (to mimic the bitter metallic taste of SDF) was painted onto all exposed tooth root surfaces using a small disposable brush. This procedure will be repeated after 12 and 24 months.In addition, instructions on oral hygiene (OHI) tailored to the individual's condition was given, and a tube of toothpaste containing 1,000 ppm fluoride (the most popular type of adult toothpaste in the Hong Kong market) was provided. The OHI and provision of toothpaste will be repeated at 6-month intervals.
  Interventions: Other: water as placebo
- silver diammine fluoride (Experimental): the subjects received the same intervention as those provided to subjects in the control group except that a 38% SDF solution (Saforide, Toyo Seiyaku Kasei Co. Ltd, Osaka, Japan) instead of the placebo solution was painted onto the exposed tooth root surfaces. This treatment was repeated after 12 and 24 months.
  Interventions: Drug: silver diammine fluoride

INTERVENTIONS:
Other: water as placebo — topical application of water as a placebo in the control arm
  Other Names: water
  Arms: control
Drug: silver diammine fluoride — topical application of the SDF solution onto tooth root surfaces
  Other Names: SDF
  Arms: silver diammine fluoride

SUMMARY:
This study was a randomized clinical trial lasting for 24 months in two study sites, Hong Kong (water fluoridated) and Guangzhou (non-fluoridated area). A total of 534 subjects will be recruited from elderly social centers located in different districts in the two study sites (260 & 274). Baseline clinical examination was conducted by a single calibrated examiner in the social centers using an intra-oral LED light, mouth mirrors and probes. Subjects were randomly allocated into two study groups and receive interventions accordingly. Follow-up examinations at 6-month intervals were carried out to assess the clinical outcomes, i.e. whether new root caries developed and whether the active root caries found at baseline become arrested. Results of this study could provide the much needed evidence to guide the dental professionals in Hong Kong and China, and possibly worldwide in deciding on the most appropriate intervention for the prevention and management of this common dental disease of the older adults.

DETAILED DESCRIPTION:
The primary and secondary outcome of this study was new root caries and arrested root caries. A root surface with new caries experience was recorded when a root surface which was sound at baseline was found to have a carious lesion or a filling at a follow-up examination. Arrested root caries was recorded when the active root caries found at baseline changed into inactive root caries at follow-up. The status of each root surface was recorded using the codes recommended by the International Caries Detection and Assessment System (ICDAS Ⅱ) Coordinating Committee in 2009.

A mean root caries increment of around 0.8 root surface per year of control group was reported in a previous clinical trial conducted in Hong Kong. Thus, in this study, a 24-month increment of 1.6 new decayed root surfaces and a standard deviation of 2 was anticipated. In order to show that a 50% difference in mean caries increment between the test and control groups was statistically significant using a 2-sample t-test at a 5% significance level and at an 80% power, a sample size of 100 subjects in each group was required. Allowing for a drop-out rate of 20% over 24 months, a total of 480 subjects (120 in each group each site) were needed.

ELIGIBILITY:
Inclusion Criteria:

1. have at least 5 teeth with exposed root surfaces and not indicated for extraction, and
2. living in the community and have self-care ability for normal daily activities.

Exclusion Criteria:

1. have life-threatening or serious health problems,
2. have cognitive problems in communication or in receiving oral hygiene instructions
3. have salivary gland diseases or received radiotherapy in the head and neck region.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Tooth Root Caries Lesions | 24 months
  Tooth roots that have changed from sound at baseline to decayed at the evaluation examination will be counted in the clinical examination

SECONDARY OUTCOMES:
Arrested root caries lesions | 24 months
  Active tooth root caries lesions at baseline that has changed to inactive root caries lesions at the evaluation examination

CONTACTS AND LOCATIONS:
Overall Officials: Edward CM Lo, BDS, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- China (2):
  - Sun Yat-sen University, Guangzhou, Guangdong
  - The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Will consider individual request case by case